CLINICAL TRIAL: NCT03076034
Title: Utility of Cortical Bone Tissue Properties in the Assessment of Fracture Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tamara Rozental, Associate Professor, Harvard Medical School, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014P000226
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Distal Radius Fracture; Osteoporosis; Hip Fractures
MeSH Terms: conditions — Wrist Fractures; Osteoporosis; Hip Fractures

STUDY DESIGN:
Intervention Model Description: Observational
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Post-menopausal women (Experimental): We will use the handheld Osteoprobe device to measure cortical bone reference point indentation properties.
  Interventions: Device: Reference Point Indentation
- Males over 50 years (Experimental): We will recruit males to this second study arm, to use the handheld Osteoprobe device to measure cortical bone reference point indentation properties.
  Interventions: Device: Reference Point Indentation

INTERVENTIONS:
Device: Reference Point Indentation — The "Osteoprobe": Since these first reports of indentation measurements in humans in vivo, a more 'user-friendly' device, the Osteoprobe® has been developed by Active Life Scientific (Santa Barbara, CA) (10). The Osteoprobe®, which we will use in the current study, is smaller than the previous reference point indentation (RPI) instrument and is designed to be used in a hand-held fashion to allow for rapid measurements. The new instrument does not require a reference probe, because the inertia of the instrument keeps it adequately fixed in space during the short time of the indentation impact (~0.25 milliseconds). The main parameter measured is the distance that the probe further indents into the bone from the reference point. Key components of the Osteoprobe® include an impact generation mechanism, a displacement transducer, and a probe made of hardened stainless steel with a 90 degree conical tip, with a tip diameter of ~375 µm.
  Other Names: Osteoprobe

SUMMARY:
The objective of this study is to determine whether a new minimally invasive method for in vivo measurement of cortical bone tissue properties can identify those who are at risk for fragility fractures of the hip and radius. The investigators hypothesis is that women with fragility fractures of the hip and radius have altered cortical bone tissue properties compared to non-fracture controls independent of standard clinical tests, such as bone mineral density (BMD) by dual-energy x-ray absorptiometry (DXA).

DETAILED DESCRIPTION:
The objective of this study is to determine whether a new minimally invasive method for in vivo measurement of cortical bone tissue properties can identify those who are at risk for fragility fractures of the hip and radius. The investigators hypothesis is that women with fragility fractures of the hip and radius have altered cortical bone tissue properties compared to non-fracture controls independent of standard clinical tests, such as BMD. To test these hypotheses, The investigators propose two aims:

Aim 1: Compare cortical bone tissue properties as assessed in vivo by reference point indentation in women with hip fractures and non-fracture controls.

The investigators will compare cortical bone tissue material properties, as assessed by novel in vivo indentation at the mid-tibia in postmenopausal women with recent hip fractures (n) and age-similar controls without fractures (n=). In addition to in vivo indentation measurements, The investigators will assess hip and spine BMD by DXA; as well as other factors that may influence risk of fractures (e.g, vit D status, medication use and physical activity). Hypotheses: Postmenopausal women with hip fractures will have worse bone tissue material properties compared to non-fracture controls even after adjustment for BMD and other potential confounders.

Aim 2: Compare cortical bone tissue properties as assessed in vivo by reference point indentation in women with distal radius fractures to non-fracture controls.

The investigators will compare cortical bone tissue material properties, as assessed by novel in vivo indentation at the mid-tibia in postmenopausal women with recent distal radius fractures (n) and age-similar controls without fractures (n=). In addition to in vivo indentation measurements, The investigators will assess hip and spine BMD by DXA; as well as other factors that may influence risk of fractures (e.g, vit D status, medication use and physical activity). Hypotheses: Postmenopausal women with distal radius fractures will have worse bone tissue material properties compared to non-fracture controls even after adjustment for BMD and other potential confounders.

Successful completion of this project will address the need to better assess bone mechanical properties at the tissue level in order to accurately predict fracture risk. The study will provide novel information about possible clinical utility of minimally invasive, in vivo bone indentation measurements to measure bone strength and its relationship to fracture risk.

Aim 3: An amendment to the protocol expanded the study population to now include males >50 years who present with distal radius fractures and those who present for a reason other than fracture (non-fracture controls). Hypotheses: Men >50 years with distal radius fractures will have worse bone tissue material properties compared to non-fracture controls even after adjustment for BMD and other potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Women with hip and wrist fractures within 2 weeks of presentation
* Non-fracture controls

Exclusion Criteria:

* Unable to undergo BMD by DXA or high-resolution peripheral quantitative computed tomography (HR-pQCT)
* History of skeletal metastasis, primary hyperparathyroidism, Paget's disease, multiple myeloma
* Treatment with bisphosphonate, estrogen (within previous 3 years), teriparatide therapy, calcitonin, selective estrogen receptor modulator (SERMs,within previous 3 years)
* Use of glucocorticoids continuously for more than 3 months, use of anticonvulsants
* Prior fracture in adulthood (>age 18) for healthy controls

Amendment to protocol added Arm 2, to include males >50 years with otherwise similar eligibility criteria.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2015-01-26 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Cortical bone tissue properties by reference point indentation | Day 1
  Osteoprobe measurement
Bone mineral density (BMD) by dual-energy x-ray absorptiometry (DXA) | Day 1
  DXA at the hip and spine

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Rozental, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03076034/ICF_000.pdf